CLINICAL TRIAL: NCT03190265
Title: A Randomized Phase 2 Study of the Safety, Efficacy, and Immune Response of CRS-207, Nivolumab, and Ipilimumab With or Without GVAX Pancreas Vaccine (With Cyclophosphamide) in Patients With Previously Treated Metastatic Pancreatic Adenocarcinoma
Brief Title: Study of CRS-207, Nivolumab, and Ipilimumab With or Without GVAX Pancreas Vaccine (With Cy) in Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Aduro Biotech, Inc. (Industry); Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1790; IRB00137389 (Other: Johns Hopkins University); 5P01CA247886-02 (NIH)
Record Dates: First submitted 2017-06-15; First posted 2017-06-16 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer
Keywords: CY; Cyclophosphamide; Pancreatic Vaccine; GVAX; Nivolumab; Vaccine; Ipilimumab; CRS-207; Immunotherapy; PD-1; Adenocarcinoma; Carcinoma; Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Carcinoma; Neoplasms | interventions — Cyclophosphamide; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: CY, Nivolumab, Ipilimumab, GVAX, CRS-207 (Experimental)
  Interventions: Drug: Cyclophosphamide; Drug: Nivolumab; Drug: Ipilimumab; Drug: GVAX Pancreas Vaccine; Drug: CRS-207
- Arm B: Nivolumab, Ipilimumab, CRS-207 (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: CRS-207

INTERVENTIONS:
Drug: Cyclophosphamide — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Cyclophosphamide (200 mg/m2) will be administered IV on day 1 of Cycles 1 and 2.
  Other Names: CY
  Arms: Arm A: CY, Nivolumab, Ipilimumab, GVAX, CRS-207
Drug: Nivolumab — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Nivolumab (360 mg) will be administered IV on day 1 of Cycles 1-6.
  Other Names: anti-PD-1, OPDIVO
Drug: Ipilimumab — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Ipilimumab (1 mg/kg) will be administered IV on Day 1 of Cycles 1, 3, and 5.
  Other Names: YERVOY®
Drug: GVAX Pancreas Vaccine — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Vaccine will be administered on Day 2 of Cycles 1 and 2.
  Other Names: GVAX, PANC 10.05 pcDNA-1/GM-Neo and PANC 6.03 pcDNA-1/GM-Neo vaccine
  Arms: Arm A: CY, Nivolumab, Ipilimumab, GVAX, CRS-207
Drug: CRS-207 — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 (1 × 109 CFU) will be administered IV on Day 2 of Cycles 3-6.
  Arms: Arm A: CY, Nivolumab, Ipilimumab, GVAX, CRS-207
Drug: CRS-207 — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 (1 × 109 CFU) will be administered IV on Day 2 of Cycles 1-6.
  Arms: Arm B: Nivolumab, Ipilimumab, CRS-207

SUMMARY:
The purpose of this study is to study the safety and clinical activity of nivolumab and ipilimumab in combination with either sequential administration of CY/GVAX pancreas vaccine followed by CRS-207 (Arm A) or with administration of CRS-207 alone (Arm B) in patients with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Have histologically or cytologically proven adenocarcinoma of the pancreas.
3. Have metastatic disease.
4. Have disease progression.
5. Patients with the presence of at least one measurable lesion.
6. Patient's acceptance to have a tumor biopsy of an accessible lesion at baseline and on treatment if the lesion can be biopsied with acceptable clinical risk (as judged by the investigator).
7. ECOG performance status 0 or 1
8. Life expectancy of greater than 3 months.
9. Patients must have adequate organ and marrow function defined by study-specified laboratory tests.
10. Must use acceptable form of birth control while on study.
11. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Known history or evidence of brain metastases.
2. Had surgery within the last 28 days
3. Had chemotherapy, radiation, or biological cancer therapy within the last 14 days
4. Have received a prophylactic vaccine within 14 days or received a live vaccine within 30 days of planned start of study therapy.
5. Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2,or anti-CTLA4
6. Systemic steroids within the last 14 days
7. Use more than 2 g/day of acetaminophen.
8. Patients on immunosuppressive agents.
9. Patients receiving growth factors within the last 14 days
10. Known allergy to both penicillin and sulfa.
11. Severe hypersensitivity reaction to any monoclonal antibody.
12. Have artificial joints or implants that cannot be easily removed
13. Have any evidence of clinical or radiographic ascites.
14. Have significant and/or malignant pleural effusion
15. Have had a new pulmonary embolism, extremity deep venous thromboembolism, or portal vein thrombosis within 2 months of study treatment
16. Infection with HIV or hepatitis B or C at screening
17. Significant heart disease
18. Conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures
19. Are pregnant or breastfeeding.
20. Have rapidly progressing disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2023-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins SKCCC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: CY, Nivolumab, Ipilimumab, Pancreas GVAX, CRS-207: Cyclophosphamide: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Cyclophosphamide (200 mg/m2) will be administered IV on day 1 of Cycles 1 and 2.
  Nivolumab: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Nivolumab (360 mg) will be administered IV on day 1 of Cycles 1-6.
  Ipilimumab: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Ipilimumab (1 mg/kg) will be administered IV on Day 1 of Cycles 1, 3, and 5.
  GVAX Pancreas Vaccine: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Vaccine will be administered on Day 2 of Cycles 1 and 2.
  CRS-207: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 (1 × 109 CFU) will be administered IV on Day 2 of Cycles 3-6.
Period: Overall Study
Arm/Group | Arm A: CY, Nivolumab, Ipilimumab, Pancreas GVAX, CRS-207 | Arm B: Nivolumab, Ipilimumab, CRS-207
Started | 31 | 30
Completed | 11 | 8
Not Completed | 20 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: CY, Nivolumab, Ipilimumab, GVAX, CRS-207 | Arm B: Nivolumab, Ipilimumab, CRS-207 | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 20 | 34
  >=65 years | 17 | 10 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 18 | 16 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 31 | 28 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 27 | 28 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Using Response Evaluation Criteria for Solid Tumors (RECIST 1.1)
Description: Objective Response Rate (ORR) is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions. Participants who discontinue due to toxicity or clinical progression prior to post-baseline tumor assessments will be considered as non-responders. Participants who discontinue for other reasons prior to their first dose of study drug will not included in the analysis.
Time Frame: 18 months
Population: Only 29/30 participants in Arm A were evaluable for this endpoint. One participant was not evaluable after they discontinued prior to their first scan for a reason other than toxicity or progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: CY, Nivolumab, Ipilimumab, Pancreas GVAX, CRS-207 | Arm B: Nivolumab, Ipilimumab, CRS-207
Number analyzed (Participants) | 29 | 27
Participants | 0 | 2

2. Secondary Outcome: Number of Participants Experiencing Grade 3 or Above Study Drug-related Adverse Events (AEs)
Description: When calculating the incidence of AEs, each AE (as defined by NCI CTCAE v4.03) will be counted only once for a given subject. Laboratory abnormalities that were asymptomatic and not clinically significant were excluded.
Time Frame: 21 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: CY, Nivolumab, Ipilimumab, Pancreas GVAX, CRS-207 | Arm B: Nivolumab, Ipilimumab, CRS-207
Number analyzed (Participants) | 30 | 27
Participants | 10 | 10

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were evaluated for up to 21 months. All-cause mortality was evaluated for up to 30 months. During the survival follow-up portion of the trial, patients in both Arms A and B were evaluated for all-cause mortality past the time frame for treatment and the assessment of adverse events.
Description: Only 30 participants in Arm A and 27 participants in Arm B were assessed for Serious and Other (Not Including Serious) Adverse Events. Four participants were withdrawn prior to their first dose of study drug (1 in Arm A and 3 in Arm B) and were therefore not assessed for Serious and Other (Not Including Serious) Adverse Events.
Arm/Group | Arm A: CY, Nivolumab, Ipilimumab, Pancreas GVAX, CRS-207 | Arm B: Nivolumab, Ipilimumab, CRS-207
All-Cause Mortality (participants affected / at risk) | 28/30 | 27/27
Serious Adverse Events (participants affected / at risk) | 24/30 | 21/27
Other Adverse Events (participants affected / at risk) | 30/30 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: CY, Nivolumab, Ipilimumab, Pancreas GVAX, CRS-207 (N=30) | Arm B: Nivolumab, Ipilimumab, CRS-207 (N=27)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 1 (2)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 3 (3)
Biliary tract infection (Infections and infestations) | 2 (2) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Disease progression (General disorders) | 13 (13) | 14 (14)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Embolic or Cardiovascular Event (Cardiac disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal sticture (Gastrointestinal disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GI tube site bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Immune Thrombocytopenia Purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Listeria monocytogenes bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Lower GI Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Radiculitis (Nervous system disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 5 (5)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)
Thyroiditis (Endocrine disorders) | 2 (2) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: CY, Nivolumab, Ipilimumab, Pancreas GVAX, CRS-207 (N=30) | Arm B: Nivolumab, Ipilimumab, CRS-207 (N=27)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 13 (17) | 13 (17)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (6) | 5 (5)
Alkaline phosphatase increased (Investigations) | 5 (5) | 5 (8)
Anemia (Blood and lymphatic system disorders) | 10 (16) | 3 (5)
Anorexia (Gastrointestinal disorders) | 13 (14) | 10 (11)
Anxiety (Psychiatric disorders) | 5 (5) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 5 (7)
Ascites (Gastrointestinal disorders) | 4 (5) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (14)
Biliary stricture (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 4 (4)
Blood bilirubin increased (Investigations) | 4 (6) | 2 (2)
Blurred vision (Eye disorders) | 2 (2) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Chest pain (Cardiac disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 17 (41) | 26 (80)
Constipation (Gastrointestinal disorders) | 8 (11) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 7 (13) | 9 (19)
Dizziness (Nervous system disorders) | 4 (4) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Edema limbs (General disorders) | 7 (10) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fatigue (General disorders) | 13 (19) | 12 (16)
Fever (General disorders) | 18 (44) | 24 (120)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 5 (7) | 7 (22)
Hematoma (Vascular disorders) | 0 (0) | 3 (3)
Hematuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (5) | 2 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 6 (6)
Hypertension (Vascular disorders) | 12 (39) | 16 (50)
Hyperthyroidism (Endocrine disorders) | 3 (4) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 7 (15) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 5 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (10) | 2 (2)
Hypotension (Vascular disorders) | 9 (22) | 16 (36)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3)
Localized edema (General disorders) | 2 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 13 (23) | 22 (44)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0)
Mucositis oral (Infections and infestations) | 3 (3) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (14)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 16 (29) | 12 (22)
Non-cardiac chest pain (General disorders) | 2 (3) | 1 (1)
Pain (General disorders) | 4 (5) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 8 (9) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 9 (11) | 4 (6)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 8 (28) | 5 (18)
Sinus tachycardia (Cardiac disorders) | 19 (43) | 19 (58)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 4 (5)
Thromboembolic event (Vascular disorders) | 4 (5) | 2 (2)
Thrush (Infections and infestations) | 5 (5) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (4) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Vaccine site adminstration discomfort (Skin and subcutaneous tissue disorders) | 16 (28) | 0 (0)
Vaccine site erythema (Skin and subcutaneous tissue disorders) | 26 (51) | 0 (0)
Vaccine site induration (Skin and subcutaneous tissue disorders) | 26 (47) | 0 (0)
Vaccine site pain (Skin and subcutaneous tissue disorders) | 14 (18) | 0 (0)
Vaccine site pruritis (Skin and subcutaneous tissue disorders) | 26 (44) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (15) | 9 (13)
Weight gain (Investigations) | 2 (2) | 2 (2)
Weight loss (Investigations) | 19 (31) | 16 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT03190265/Prot_SAP_000.pdf